CLINICAL TRIAL: NCT05478655
Title: Predictors of Treatment Failure Pain Among Patients With Mine-explosive Wounds
Acronym: PTFPAPM-EW
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Vasyl' Horoshko, Chief researcher, Bogomolets National Medical University
Other Study IDs: №158 23/05/2022
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain
Keywords: Chronic pain, mine-explosive wounds
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective analysis: A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation In all patients, the assessment of anesthetic risk was carried out according to the ASA scale.The basic tool for pain intensity research was a visual analog scale.The study of the neuropathic component of pain was carried out using the diagnostic questionnaire for the detection of neuropathic pain Didier Bouhassiraa, Nadine Attala et al. Pain, 2005, 114: 29-36. Study of the presence of an acute stress reaction scale The Hospital Anxiety and Depression Scale. The presence of post-traumatic stress disorders was studied using the Mississippi scale of post-traumatic stress disorders (military version). Satisfaction with the results of treatment was studied using the Chaban Quality of Life Scale.
  Interventions: Other: visual analog scale
- prospective study: Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022. Data collection was carried out during the Russian invasion of Ukraine and the offensive on Kyiv. All patients with gunshot wounds were evacuated to the stage of treatment - the National Military Medical Clinical Center "Main Military Clinical Hospital". The research was conducted using the same methods as during the retrospective analysis. The exception was the study period during treatment at the military medical clinical center: here it was 14 days.
  Interventions: Other: visual analog scale

INTERVENTIONS:
Other: visual analog scale — VAS was studied: 1) before and after anesthesia - at the stage of the medical and nursing brigade, military mobile hospital, military medical clinical center; 2) at the stage of the medical and nursing team - within 2 days; 3) at the stage of the military mobile hospital - within 5 days; 4) at the stage of the military medical clinical center - within 7 days, at the time of discharge from the hospital and further 1, 3, 6, 12 months after the injury; 5) at the rehabilitation stage. Intervals between analgesia were also studied.
  Other Names: neuropathic pain Didier Bouhassiraa, Nadine Attala et al. Pain, 2005, 114: 29-36 (DN4).; ASA; The Hospital Anxiety and Depression Scale; Mississippi PTSD scale (military version); Chaban Quality of Life Scale

SUMMARY:
Mine-explosive wounds in the general structure of combat sanitary losses reach 25%. They are characterized by significant damage resulting in high intensity pain. In patients who received mine-explosive injuries in the conditions of hostilities, such pain has its own unique features. It is necessary to pay more attention to the problem of pain treatment in patients of this category, because about 87.2% of cases have negative results of treatment - it becomes chronic.

DETAILED DESCRIPTION:
The peculiarities of pain in patients with mine-explosive wounds depending on the localization of the wound at the stages of treatment need to be studied, because the subjective feelings and emotional experiences experienced by patients during the wounding in combat conditions through the prism of psychological disorders have their own characteristics. Since in 87.2% of cases it is not possible to achieve a positive result of treatment, the data of our study will play an important role in their treatment.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain, mine-explosive wounds

Exclusion Criteria:

* absence of mine-explosive wounds

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study was carried out on the basis of the National Military Medical Clinical Center "Main Military Clinical Hospital". All patients participated in Operation Joint Forces and received gunshot wounds during combat operations.
  A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022. Data collection was carried out during the Russian invasion of Ukraine and the offensive on Kyiv.
Sampling Method: Non-Probability Sample
Enrollment: 1166 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 12 months
  evaluation of the number of points
Didier Bouhassiraa DN4 | 12 months
  evaluation of the number of points
The Hospital Anxiety and Depression Scale | 12 months
  evaluation of the number of points
Chaban Quality of Life Scale | 12 months
  evaluation of the number of points

CONTACTS AND LOCATIONS:
Locations (1):
- Bogomolets National Medical University, Ministry of Health of Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided
I plan to share